CLINICAL TRIAL: NCT05331001
Title: Quality of Care in Centers Providing Extracorporeal Membrane Oxygenation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Tharusan Thevathasan, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ECMO Quality of Care
Record Dates: First submitted 2022-04-10; First posted 2022-04-15 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Cardiogenic Shock; Myocardial Infarction; Cardiac Arrest; Extracorporeal Circulation; Complications
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical doctors: Medical doctors who are employed as permanent staff in a cardiac arrest center which provides extracorporeal membrane oxygenation.
- Nurses: Nurses who are employed as permanent staff in a cardiac arrest center which provides extracorporeal membrane oxygenation.

SUMMARY:
Cardiac arrest centers are specialized in treating critically ill patients with severe cardiovascular diseases, such as cardiac arrest, cardiogenic shock or acute myocardial infarction. Diagnostic and therapeutic measures, such as the use of devices for extracorporeal life support, require highly specialized training and skills. Apart from extensive medical expertise, physicians and nurses may be exposed to exceptional levels of occupational stressors. Therefore, excellent medical, psychological and inter-personal training of the medical staff is essential to improve patient outcomes. Assessment of quality of care is important to provide continuous improvement in patient care and team performance. To the best of our knowledge, there is no study which examined the quality of care in cardiac arrest centers across key dimensions of quality of care. Therefore, we aim to assess a bundle of key dimensions, that is psychological strain (P), resource utilization (R), interaction (I) between doctoral and nursing staff, costs of care (C) and education (E) programs for staff (PRICE scheme). A cross-sectional study will be conducted with doctors and nurses, using a digital quesitonnaire that will cover the five dimensions of the PRICE scheme.

ELIGIBILITY:
Inclusion Criteria:

* Adult medical doctors or nurses
* Permament staff in the cardiac arrest center
* Cardiac arrest center that provides therapy with extracorporeal membrane oxygenation (ECMO)

Exclusion Criteria:

* No permanent employment in a cardiac arrest center
* Non-adult staff
* Not a medical doctor or nurse
* Cardiac arrest center that does not provide therapy with ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Permament adult staff which is employed in a cardiac arrest center that provides therapy with extracorporeal membrane oxygenation (ECMO). Medical doctors and nurses are included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Psychological strain (P) | During one week all permanent staff of a cardiac arrest center will be asked to fill out the standardized questionnaire.
  The psychologial strain of permanent staff in the cardiac arrest center will be assessed based on a standardized questionnaire.

SECONDARY OUTCOMES:
Ressource utilization (R) | During one week all permanent staff of a cardiac arrest center will be asked to fill out the standardized questionnaire.
  The availability of material and non-material ressources and the extent of ressource utilization in the cardiac arrest center will be assessed based on a standardized questionnaire.
Interaction (I) | During one week all permanent staff of a cardiac arrest center will be asked to fill out the standardized questionnaire.
  The quality of inter-professional interactions between medical doctors and nurses in the cardiac arrest center will be assessed based on a standardized questionnaire.
Costs (C) of care | During one week all permanent staff of a cardiac arrest center will be asked to fill out the standardized questionnaire.
  The costs of care in the cardiac arrest center will be assessed based on a standardized questionnaire.
Education (E) programs | During one week all permanent staff of a cardiac arrest center will be asked to fill out the standardized questionnaire.
  The availability and quality of education programs in the cardiac arrest center will be assessed based on a standardized questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Skurk, MD, Study Director — Charite University; Tharusan Thevathasan, MD, Principal Investigator — Charite University

IPD SHARING:
Plan to Share IPD: No